CLINICAL TRIAL: NCT02382939
Title: A Multicentre, Multinational, Randomised, Open-labelled, Parallel-group, Active-controlled Trial to Compare the Safety of Once Weekly Dosing of Somapacitan With Daily Norditropin® FlexPro® for 26 Weeks in Previously Human Growth Hormone Treated Adults With Growth Hormone Deficiency
Brief Title: A Trial to Compare the Safety of Once Weekly Dosing of Somapacitan With Daily Norditropin® FlexPro® for 26 Weeks in Previously Human Growth Hormone Treated Adults With Growth Hormone Deficiency
Acronym: REAL 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-4043; 2014-000290-39 (EudraCT Number); U1111-1152-3664 (Other: WHO); JapicCTI-152850 (Other: JAPIC)
Record Dates: First submitted 2015-02-10; First posted 2015-03-09 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Adult Growth Hormone Deficiency; Growth Hormone Disorder
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somapacitan; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- somapacitan (Experimental)
  Interventions: Drug: somapacitan
- hGH (somatropin) (Active Comparator)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somapacitan — Administered subcutaneously (s.c., under the skin) with an investigational pen once weekly for a 26 week period (8 weeks' dose titration, 18 weeks' fixed dose treatment) followed by 1 week washout.
  Arms: somapacitan
Drug: somatropin — Administered subcutaneously (s.c., under the skin) with a prefilled pen (Norditropin® FlexPro®) daily for a 26 week period (8 weeks' dose titration, 18 weeks' fixed dose treatment) followed by 1 week washout.
  Arms: hGH (somatropin)

SUMMARY:
This trial is conducted in Europe and Asia. The aim of the trial is to compare the safety of once weekly dosing of somapacitan (administered with an investigational pen) with daily Norditropin® FlexPro® (somatropin delivered within a prefilled pen) for 26 weeks in previously human growth hormone (hGH) treated adults with growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria: - Male or female of at least 18 years of age and not more than 79 years of age at the time of signing informed consent - Adult growth hormone deficiency diagnosed for 6 months or longer (defined as 180 days) prior to screening - Treatment with hGH (human growth hormone) for at least 6 months at screening - If applicable, hormone replacement therapies for any other hormone deficiencies, adequate and stable for at least 90 days prior to randomisation as judged by the investigator Exclusion Criteria: - Active malignant disease or history of malignancy. Exceptions to this exclusion criterion: Resected in situ carcinoma of the cervix and squamous cell or basal cell carcinoma of the skin with complete local excision. / Subjects with GHD (growth hormone deficiency) attributed to treatment of intracranial malignant tumours or leukaemia, provided that a recurrence-free survival period of at least 5 years is documented in the subject's file - For patients with surgical removal or debulking of pituitary adenoma or other benign intracranial tumour within the last 5 years: Evidence of growth of pituitary adenoma or other benign intracranial tumour within the last 12 months (defined as below or equal to 365 days) before randomisation. Absence of growth must be documented by two post-surgery MRI or CT scans. The most recent MRI or CT scan must be performed below or equal to 9 months (defined as below or equal to 270 days) prior to randomisation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2016-01-04 (Actual); Study Completion 2016-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (27):
- Denmark (3):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, København Ø
  - Novo Nordisk Investigational Site, Odense
- France (5):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Dijon
  - Novo Nordisk Investigational Site, Saint-Herblain
- Germany (3):
  - Novo Nordisk Investigational Site, Aachen
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Frankfurt
- Japan (8):
  - Novo Nordisk Investigational Site, Bunkyo-ku, Tokyo
  - Novo Nordisk Investigational Site, Itabashi-ku, Tokyo
  - Novo Nordisk Investigational Site, Izumo, Shimane
  - Novo Nordisk Investigational Site, Kobe, Hyogo
  - Novo Nordisk Investigational Site, Kobe-shi, Hyogo
  - Novo Nordisk Investigational Site, Kyoto-shi Kyoto
  - Novo Nordisk Investigational Site, Okayama, Okayama
  - Novo Nordisk Investigational Site, Sagamihara-shi, Kanagawa
- Sweden (3):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Stockholm
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Exeter
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester

REFERENCES:
- [Derived] Takahashi Y, Biller BMK, Fukuoka H, Ho KKY, Rasmussen MH, Nedjatian N, Svaerke C, Yuen KCJ, Johannsson G. Weekly somapacitan had no adverse effects on glucose metabolism in adults with growth hormone deficiency. Pituitary. 2023 Feb;26(1):57-72. doi: 10.1007/s11102-022-01283-3. Epub 2022 Nov 15. PMID 36380045
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 26 sites in 6 countries. All 26 sites screened and randomised/ assigned patients to treatment. Denmark: 3 sites; France: 5 sites; Germany: 3 sites; Sweden: 3 sites; United Kingdom: 5 sites; Japan: 7 sites.
Pre-assignment Details: Participants, who were diagnosed with adults with growth hormone deficiency ≥ 6 months (defined as 180 days) prior to screening and receiving treatment with human growth hormone at least 6 months (defined as 180 days) at screening, were enrolled.
Groups:
- Norditropin: Participants received subcutaneous (s.c.) injections of Norditropin daily for 26 weeks (8 weeks dose titration followed by 18 weeks fixed dose treatment) followed by 1 week washout. The starting dose of Norditropin was 0.2 mg/day (except females on oral oestrogen: 0.3 mg/day; participants older than 60 years: 0.1 mg/day). An individualised dose titration regimen was used. Adjustment of dose was performed at weeks 2, 4, 6 and 8 based on insulin-like growth factor-I standard deviation score (IGF-I SDS) values:
  IGF-I SDS > 3: dose reduction by 0.1 mg/day 2 < IGF-I SDS ≤ 3: dose reduction by 0.05 mg/day 0 < IGF-I SDS ≤ 2: No need of dose adjustment
  * 2 < IGF-I SDS ≤ 0: Dose increment by 0.1 mg/day IGF-I SDS ≤ -2: Dose increment by 0.2 mg/day After the last dose adjustment (if any) at week 8, the individual dose level was fixed. The minimum and maximum daily dose was set to 0.05 mg and 1.1 mg (Japan: maximum daily dose was 1.0 mg).
- Somapacitan: Participants received s.c. injections of somapacitan once-weekly for 26 weeks (8 weeks dose titration followed by 18 weeks fixed dose treatment) followed by 1 week washout. The starting dose of somapacitan was 1.5 mg/week (except females on oral oestrogen 2.0 mg/week; participants older than 60 years 1.0 mg/week). An individualised dose titration regimen was used. Adjustment of dose was performed at weeks 2, 4, 6 and 8 based on IGF-I SDS values:
  IGF-I SDS > 3: dose reduction by 1 mg 2 < IGF-I SDS ≤ 3: dose reduction by 0.5 mg 0 < IGF-I SDS ≤ 2: No need for dose adjustment
  * 2 < IGF-I SDS ≤ 0: Dose Increment by 0.7 mg IGF-I SDS ≤ -2: Dose Increment by 1.5 mg After the last dose adjustment (if any) at week 8, the individual dose level was fixed. The minimum and maximum weekly dose was set to 0.1 mg and 8 mg.
Period: Overall Study
Arm/Group | Norditropin | Somapacitan
Started | 31 | 61
Exposed | 31 | 61
Completed | 28 | 58
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all randomised participants that received at least one dose of randomised treatment.
Groups:
- Norditropin: Participants received s.c. injections of Norditropin daily for 26 weeks (8 weeks dose titration followed by 18 weeks fixed dose treatment) followed by 1 week washout. The starting dose of Norditropin was 0.2 mg/day (except females on oral oestrogen: 0.3 mg/day; participants older than 60 years: 0.1 mg/day). An individualised dose titration regimen was used. Adjustment of dose was performed at weeks 2, 4, 6 and 8 based on IGF-I SDS values:
  IGF-I SDS > 3: dose reduction by 0.1 mg/day 2 < IGF-I SDS ≤ 3: dose reduction by 0.05 mg/day 0 < IGF-I SDS ≤ 2: No need of dose adjustment
  * 2 < IGF-I SDS ≤ 0: Dose increment by 0.1 mg/day IGF-I SDS ≤ -2: Dose increment by 0.2 mg/day After the last dose adjustment (if any) at week 8, the individual dose level was fixed. The minimum and maximum daily dose was set to 0.05 mg and 1.1 mg (Japan: maximum daily dose was 1.0 mg).
- Total: Total of all reporting groups
Arm/Group | Norditropin | Somapacitan | Total
Number analyzed (Participants) | 31 | 61 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (17.1) | 48.1 (16.2) | 49.3 (16.5)
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 23 | 50 | 73
  ≥65 years | 8 | 11 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 28 | 42
  Male | 17 | 33 | 50

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: An adverse event can be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. Presented results are event rate per 100 patient years of exposure.
Time Frame: Weeks 0 - 26
Population: Safety analysis set: all randomised participants that received at least one dose of randomised treatment.
Measure: Number; unit: Events per 100 patient years
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 31 | 61
Events per 100 patient years | 530.8 | 514.2

2. Primary Outcome: Incidence of Injection Site Reactions
Description: Presented results are event (injection site reaction) rate per 100 patient years of exposure.
Time Frame: Weeks 0- 26
Population: Safety analysis set: all randomised participants that received at least one dose of randomised treatment.
Measure: Number; unit: Events per 100 patient years
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 31 | 61
Events per 100 patient years | 0 | 6.5

3. Secondary Outcome: Occurrence of Anti-NNC0195-0092 Antibodies
Description: Number of participants with anti-somapacitan (NNC0195-0092) antibodies are presented.
Time Frame: At week 0 (baseline), and at week 2, 4, 8, 16, 25 and 27
Population: Overall Number of Participants Analyzed = safety analysis set which included all randomised participants that received at least one dose of randomised treatment. Number Analyzed = number of participants with available data. This outcome measure is applicable only for the somapacitan treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Somapacitan
Number analyzed (Participants) | 61
Participants
  Week 0:: number analyzed (Participants) | 60
  Week 0: | 0
  Week 2:: number analyzed (Participants) | 60
  Week 2: | 0
  Week 4:: number analyzed (Participants) | 60
  Week 4: | 0
  Week 8:: number analyzed (Participants) | 58
  Week 8: | 0
  Week 16:: number analyzed (Participants) | 57
  Week 16: | 0
  Week 25:: number analyzed (Participants) | 60
  Week 25: | 0
  Week 27:: number analyzed (Participants) | 60
  Week 27: | 0

4. Secondary Outcome: Change in Treatment Satisfaction Questionnaire for Medication (TSQM) Scores (Effectiveness,Convenience, and Global Satisfaction Scores)
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM-9) is a psychometric measure of a patient's satisfaction with medication. It consists of 3 subscales: effectiveness, convenience and global satisfaction. Items are rated on a 5 or 7-point scale according to participants' experience with the medication. Each domain score can vary from 0 to 100 with higher scores indicating higher effectiveness of treatment, more convenient use of medication and overall greater satisfaction with the treatment.
Time Frame: Baseline (week 0), week 26
Population: Overall Number of Participants Analyzed = full analysis set which included all randomised participants that received at least one dose of randomised treatment. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 31 | 61
Score on a scale
  Effectiveness: number analyzed (Participants) | 28 | 53
  Effectiveness | 3.8 (27.4) | 9.7 (18.1)
  Convenience: number analyzed (Participants) | 28 | 55
  Convenience | 3.0 (16.5) | 15.3 (20.9)
  Global satisfaction: number analyzed (Participants) | 28 | 54
  Global satisfaction | -1.2 (15.2) | 5.4 (21.0)

ADVERSE EVENTS:
Time Frame: Baseline (week 0) to week 26.
Description: Participants in the safety analysis set contributed to the evaluation of adverse events.
Groups:
- Norditropin: Participants received s.c. injections of Norditropin daily for 26 weeks (8 weeks dose titration followed by 18 weeks fixed dose treatment) followed by 1 week washout. The starting dose of Norditropin was 0.2 mg/day (except females on oral oestrogen: 0.3 mg/day; participants older than 60 years: 0.1 mg/day). An individualised dose titration regimen was used. Adjustment of dose was performed at weeks 2, 4, 6 and 8 based on IGF-I SDS values:
  IGF-I SDS > 3: dose reduction by 0.1 mg/day 2 < IGF-I SDS ≤ 3: dose reduction by 0.05 mg/day 0 < IGF-I SDS ≤ 2: No need of dose adjustment
  * 2 < IGF-I SDS ≤ 0: Dose increment by 0.1 mg/day IGF-I SDS ≤ -2: Dose increment by 0.2 mg/day After the last dose adjustment (if any) at week 8, the individual dose level was fixed.
Arm/Group | Norditropin | Somapacitan
Serious Adverse Events (participants affected / at risk) | 2/31 | 4/61
Other Adverse Events (participants affected / at risk) | 18/31 | 30/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norditropin (N=31) | Somapacitan (N=61)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mammoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Short-bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norditropin (N=31) | Somapacitan (N=61)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Asthenia (General disorders) | 1 (1) | 4 (5)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 5 (5) | 6 (7)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (10) | 7 (11)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (11) | 12 (13)
Sciatica (Nervous system disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.